CLINICAL TRIAL: NCT02662777
Title: International, Prospective, Multicenter Registry Designed to Collect Clinical Evidence for Endoscopic Vacuum Treatment Using Eso-SPONGE® for Anastomotic Leakage After Esophageal Resection or Iatrogenic or Spontaneous Esophageal Perforation.
Brief Title: Eso-Sponge Registry
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: Universitätsklinikum Kiel (Unknown)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1317
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Leakage After Esophagectomy; Leakage After Gastrectomy; Perforation of the Esophagus
Keywords: esophageal anastomosis leakage; endoscopic vacuum therapy; esophageal perforation; upper gastrointestinal tract; esophageal leak; endoscopy
MeSH Terms: conditions — Esophageal Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eso-SPONGE® vacuum treatment: leakage after esophagectomy and gastrectomy, perforation of the esophagus
  Interventions: Device: Eso-SPONGE® vacuum treatment

INTERVENTIONS:
Device: Eso-SPONGE® vacuum treatment

SUMMARY:
This international, prospective and multicenter registry was designed to collect clinical evidence for the endoscopic vacuum treatment using Eso-SPONGE® for anastomotic leakage after esophageal resection or iatrogenic or spontaneous esophageal perforation.

DETAILED DESCRIPTION:
Anastomotic Leakages or other defects in the upper gastrointestinal tract can have serious consequences for the affected patients. Different parameters, like the size, location, time to diagnosis of the lesion, but also the general condition of the patient, have a significant influence on the clinical outcome of the patient. Often this situation is accompanied by symptoms of sepsis and a significant morbidity rate with corresponding substantial mortality rate. For this reason the treatment of this clinical situation is often a challenge for the clinician.

Besides surgical examination and the endoscopic stent system, good experiences have been obtained with the Endo-SPONGE® therapy for the lower gastrointestinal tract. In the future the endoluminal vacuum therapy for the upper gastrointestinal is available, too, with Eso-SPONGE®.

Eso-SPONGE® represent an innovative therapy concept for the treatment of this problem in the upper gastrointestinal tract, which can contribute significantly to the reduction of morbidity and mortality of the patients.

The overall success rate of endoscopic esophageal vacuum therapy in the literature ranges from 80-100%. Currently only cohort studies including a small number of patients have been performed and published. Therefore an international, prospective and multicenter registry was designed to collect clinical evidence for Eso-SPONGE treatment concept in a large population under daily clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic vacuum therapy (EVT) of anastomotic leakage after esophageal resection or spontaneous or iatrogenic perforations
* age > 18 years
* written informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anastomotic leakages after esophageal resection or gastrectomy and spontaneous or iatrogenic esophageal perforations.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Healing rate of the esophageal anastomosis leakage or esophageal perforation | until day of discharge (approximately 2 weeks)
  Reduction of the cavity, endoscopic vacuum therapy no longer necessary

SECONDARY OUTCOMES:
Number of Eso-SPONGE® changes | until day of discharge (approximately 2 weeks)
Total number of sponges used | until day of discharge (approximately 2 weeks)
  Total number of Eso-SPONGE® units used until day of discharge
Average replacement intervals | until day of discharge (approximately 2 weeks)
  Period of time between exchange of ESO-Sponge®
Duration of endoscopic vacuum therapy | until day of discharge (approximately 2 weeks)
  Number of days during which Eso-SPONGE® was applied
Complication Rate | until day of discharge (approximately 2 weeks)
  Number of Complications during endoscopic vacuum treatment (e.g. death, re-operations, stenosis, pneumonia, peritonitis, mediastinitis)

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Schafmayer, Prof. Dr., Study Chair — Universitätsklinikum Kiel
Locations (17):
- Germany (17):
  - Siloah St. Trudpert Klinikum, Pforzheim, Baden-Wurttemberg
  - Sankt Katharinen Krankenhaus, Frankfurt am Main, Hesse
  - Klinikum Herford, Herford, Hesse
  - Asklepios Klinik, Lich, Hesse
  - Klinikum Lüneburg, Klinik für Allgemein-, Viszeral- & Thoraxchirurgie, Lüneburg, Lower Saxony
  - Klinikum Wilhelmshaven, Wilhelmshaven, Lower Saxony
  - Augusta-Kliniken GmbH, Bochum, North Rhine-Westphalia
  - St. Johannes-Hospital Dortmund, Dortmund, North Rhine-Westphalia
  - EVK Herne, Herne, North Rhine-Westphalia
  - Universitätsklinikum Kiel, Kiel, Schleswig-Holstein
  - Wald-Klinikum Gera, Gera, Thuringia
  - Zentralklinik Bad Berka, Bad Berka
  - Krankenhaus der Augustinerinnen, Cologne
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Greifswald, Greifswald
  - Städtisches Krankenhaus Heinsberg, Heinsberg
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahrens M, Schulte T, Egberts J, Schafmayer C, Hampe J, Fritscher-Ravens A, Broering DC, Schniewind B. Drainage of esophageal leakage using endoscopic vacuum therapy: a prospective pilot study. Endoscopy. 2010 Sep;42(9):693-8. doi: 10.1055/s-0030-1255688. Epub 2010 Aug 30. PMID 20806153
- [Background] Bludau M, Holscher AH, Herbold T, Leers JM, Gutschow C, Fuchs H, Schroder W. Management of upper intestinal leaks using an endoscopic vacuum-assisted closure system (E-VAC). Surg Endosc. 2014 Mar;28(3):896-901. doi: 10.1007/s00464-013-3244-5. Epub 2013 Oct 23. PMID 24149851
- [Background] Brangewitz M, Voigtlander T, Helfritz FA, Lankisch TO, Winkler M, Klempnauer J, Manns MP, Schneider AS, Wedemeyer J. Endoscopic closure of esophageal intrathoracic leaks: stent versus endoscopic vacuum-assisted closure, a retrospective analysis. Endoscopy. 2013 Jun;45(6):433-8. doi: 10.1055/s-0032-1326435. Epub 2013 Jun 3. PMID 23733727
- [Background] Gubler C, Schneider PM, Bauerfeind P. Complex anastomotic leaks following esophageal resections: the new stent over sponge (SOS) approach. Dis Esophagus. 2013 Aug;26(6):598-602. doi: 10.1111/dote.12005. Epub 2012 Nov 30. PMID 23199232
- [Background] Heits N, Stapel L, Reichert B, Schafmayer C, Schniewind B, Becker T, Hampe J, Egberts JH. Endoscopic endoluminal vacuum therapy in esophageal perforation. Ann Thorac Surg. 2014 Mar;97(3):1029-35. doi: 10.1016/j.athoracsur.2013.11.014. Epub 2014 Jan 18. PMID 24444874
- [Background] Kuehn F, Schiffmann L, Rau BM, Klar E. Surgical endoscopic vacuum therapy for anastomotic leakage and perforation of the upper gastrointestinal tract. J Gastrointest Surg. 2012 Nov;16(11):2145-50. doi: 10.1007/s11605-012-2014-3. Epub 2012 Sep 5. PMID 22948839
- [Background] Lenzen H, Negm AA, Erichsen TJ, Manns MP, Wedemeyer J, Lankisch TO. Successful treatment of cervical esophageal leakage by endoscopic-vacuum assisted closure therapy. World J Gastrointest Endosc. 2013 Jul 16;5(7):340-5. doi: 10.4253/wjge.v5.i7.340. PMID 23858378
- [Background] Loske G, Schorsch T. [Endoscopic intraluminal vacuum therapy of complete esophageal-jejunal anastomotic rupture: a case report.] Viszeralmedizin. 2011; 27: 166-168.
- [Background] Loske G, Schorsch T, Muller C. Intraluminal and intracavitary vacuum therapy for esophageal leakage: a new endoscopic minimally invasive approach. Endoscopy. 2011 Jun;43(6):540-4. doi: 10.1055/s-0030-1256345. Epub 2011 Mar 29. PMID 21448855
- [Background] Loske G, Schorsch T, Müller C. Intraluminale und intracavitäre Vakuumtherapie bei Ösophagusdefekten. Z Gastroenterol. 2010; 48: 19.
- [Background] Loske G, Schorsch T, Müller C. Erste Erfahrungen mit der intraluminalen endoskopischen Vakuumschwammtherapie zur Behandlung von Duodenaldefekten. Z Gastroenterol. 2010; 48: 55
- [Background] Loske G, Schorsch T, Muller C. Endoscopic intracavitary vacuum sponge therapy of anastomotic leakage in the proximal colon after right-sided colectomy. Endoscopy. 2010;42 Suppl 2:E171-2. doi: 10.1055/s-0029-1244177. Epub 2010 Jun 16. No abstract available. PMID 20556720
- [Background] Loske G, Schorsch T, Muller C. Endoscopic intracavitary vacuum therapy of Boerhaave's syndrome: a case report. Endoscopy. 2010;42 Suppl 2:E144-5. doi: 10.1055/s-0029-1244092. Epub 2010 Apr 19. No abstract available. PMID 20405387
- [Background] Loske G, Schorsch T, Muller C. Endoscopic vacuum sponge therapy for esophageal defects. Surg Endosc. 2010 Oct;24(10):2531-5. doi: 10.1007/s00464-010-0998-x. Epub 2010 Mar 24. PMID 20333402
- [Background] Loske G, Schorsch T, Mueller CT. Endoscopic intraluminal vacuum therapy of duodenal perforation. Endoscopy. 2010;42 Suppl 2:E109. doi: 10.1055/s-0029-1243947. Epub 2010 Mar 19. No abstract available. PMID 20306395
- [Background] Loske G, Schorsch T. [Intraluminale Vakuumtherapie - ein innovativer endoskopischer Ansatz zur Therapie von duodenalen Leckagen.] Endoscopy. 2010; 23 (4). 267-269.
- [Background] Loske G, Muller C. Endoscopic vacuum-assisted closure of upper intestinal anastomotic leaks. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):601-2; author reply 602. doi: 10.1016/j.gie.2008.06.058. No abstract available. PMID 19231507
- [Background] Loske G, Muller C. [Vacuum therapy of an esophageal anastomotic leakage--a case report]. Zentralbl Chir. 2009 Jun;134(3):267-70. doi: 10.1055/s-0028-1098764. Epub 2009 Apr 22. German. PMID 19387934
- [Background] Murphy T, Jobe BA. Endoluminal management of anastomotic dehiscence after esophagectomy: an increasing quiver of options reflects the difficulty in realizing a definitive therapy. Gastrointest Endosc. 2010 Feb;71(2):387-9. doi: 10.1016/j.gie.2009.09.033. No abstract available. PMID 20152315
- [Background] Saadi A, Perentes JY, Gonzalez M, Tempia AC, Wang Y, Demartines N, Ris HB, Krueger T. Vacuum-assisted closure device: a useful tool in the management of severe intrathoracic infections. Ann Thorac Surg. 2011 May;91(5):1582-9. doi: 10.1016/j.athoracsur.2011.01.018. Epub 2011 Feb 26. PMID 21354551
- [Background] Schniewind B, Schafmayer C, Voehrs G, Egberts J, von Schoenfels W, Rose T, Kurdow R, Arlt A, Ellrichmann M, Jurgensen C, Schreiber S, Becker T, Hampe J. Endoscopic endoluminal vacuum therapy is superior to other regimens in managing anastomotic leakage after esophagectomy: a comparative retrospective study. Surg Endosc. 2013 Oct;27(10):3883-90. doi: 10.1007/s00464-013-2998-0. Epub 2013 May 25. PMID 23708716
- [Background] Schniewind B, Schafmayer C, Both M, Arlt A, Fritscher-Ravens A, Hampe J. Ingrowth and device disintegration in an intralobar abscess cavity during endosponge therapy for esophageal anastomotic leakage. Endoscopy. 2011;43 Suppl 2 UCTN:E64-5. doi: 10.1055/s-0030-1255799. Epub 2011 Feb 21. No abstract available. PMID 21341185
- [Background] Schorsch T, Muller C, Loske G. Pancreatico-gastric anastomotic insufficiency successfully treated with endoscopic vacuum therapy. Endoscopy. 2013;45 Suppl 2 UCTN:E141-2. doi: 10.1055/s-0032-1326260. Epub 2013 May 28. No abstract available. PMID 23716102
- [Background] Schorsch T, Muller C, Loske G. Endoscopic vacuum therapy of anastomotic leakage and iatrogenic perforation in the esophagus. Surg Endosc. 2013 Jun;27(6):2040-5. doi: 10.1007/s00464-012-2707-4. Epub 2012 Dec 18. PMID 23247743
- [Background] Wallstabe I, Tiedemann A, Schiefke I. Endoscopic vacuum-assisted therapy of infected pancreatic pseudocyst using a coated sponge. Endoscopy. 2012;44 Suppl 2 UCTN:E49-50. doi: 10.1055/s-0031-1291525. Epub 2012 Mar 6. No abstract available. PMID 22396274
- [Background] Wallstabe I, Tiedemann A, Schiefke I. Endoscopic vacuum-assisted therapy of an infected pancreatic pseudocyst. Endoscopy. 2011;43 Suppl 2 UCTN:E312-3. doi: 10.1055/s-0030-1256643. Epub 2011 Sep 13. No abstract available. PMID 21915843
- [Background] Wallstabe I, Plato R, Weimann A. Endoluminal vacuum therapy for anastomotic insufficiency after gastrectomy. Endoscopy. 2010;42 Suppl 2:E165-6. doi: 10.1055/s-0029-1244150. Epub 2010 Jun 16. No abstract available. PMID 20556717
- [Background] Wallstabe I, Weimann A. Eine neue endoskopische Technik im Management der Anastomoseinsuffizienz nach Ösophaguschirurgie. Z Gastroenterol 2007; 45
- [Background] Wedemeyer J, Lankisch T. [Endoscopic vacuum-assisted closure]. Internist (Berl). 2013 Mar;54(3):309-14. doi: 10.1007/s00108-012-3182-7. German. PMID 23430199
- [Background] Wedemeyer J, Schneider AS, Winkler M, Manns MP. Endoskopische Vakuumtherapie bei Perforationen und Anastomoseninsuffizienzen. Gastroenterologe. 2011; 6 (2): 120-123.
- [Background] Wedemeyer J, Brangewitz M, Kubicka S, Jackobs S, Winkler M, Neipp M, Klempnauer J, Manns MP, Schneider AS. Management of major postsurgical gastroesophageal intrathoracic leaks with an endoscopic vacuum-assisted closure system. Gastrointest Endosc. 2010 Feb;71(2):382-6. doi: 10.1016/j.gie.2009.07.011. Epub 2009 Oct 30. PMID 19879566
- [Background] Wedemeyer J, Helfritz FA, Brangewitz M, Winkler M, Manns MP, Schneider A. Endoskopische Vakuum-Schwamm-Therapie bei Leckagen im Verdauungstrakt . Gastrointest Endosc 2009; 23 (1): 41-45.
- [Background] Wedemeyer J, Schneider A, Manns MP, Jackobs S. Endoscopic vacuum-assisted closure of upper intestinal anastomotic leaks. Gastrointest Endosc. 2008 Apr;67(4):708-11. doi: 10.1016/j.gie.2007.10.064. PMID 18374029
- [Background] Weidenhagen R, Hartl WH, Gruetzner KU, Eichhorn ME, Spelsberg F, Jauch KW. Anastomotic leakage after esophageal resection: new treatment options by endoluminal vacuum therapy. Ann Thorac Surg. 2010 Nov;90(5):1674-81. doi: 10.1016/j.athoracsur.2010.07.007. PMID 20971288
- [Background] Wettstein M, Frieling T, Luthen R, Heintges T, Niederau C, Oette M, Vogt C, Vom Dahl S. [Endoscopic therapy for leaks in the gastrointestinal tract, the bile ducts and the pancreas]. Z Gastroenterol. 2011 Jun;49(6):740-8. doi: 10.1055/s-0031-1273422. Epub 2011 Jun 1. German. PMID 21638241
- [Result] Richter F, Hendricks A, Schniewind B, Hampe J, Heits N, von Schonfels W, Reichert B, Eberle K, Ellrichmann M, Baumann P, Egberts JH, Becker T, Schafmayer C. Eso-Sponge(R) for anastomotic leakage after oesophageal resection or perforation: outcomes from a national, prospective multicentre registry. BJS Open. 2022 Mar 8;6(2):zrac030. doi: 10.1093/bjsopen/zrac030. PMID 35451010